CLINICAL TRIAL: NCT04824508
Title: Effect of the Position of the Teamleader on Quality of Leadership and Team Performance
Brief Title: Position of Teamleader and Leadership Performance
Acronym: LeadPos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 4031-Sim
Record Dates: First submitted 2021-03-22; First posted 2021-04-01 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Leadership
Keywords: simulation; cardiopulmonary resuscitation; teamleader
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional position (head position) (Active Comparator): Leaderposition at the patient's head
  Interventions: Behavioral: position
- Remote position (Active Comparator): Leaderposition remote from patient and hands-off
  Interventions: Behavioral: position

INTERVENTIONS:
Behavioral: position — teamleaders are instructed to allocated position

SUMMARY:
Investigation in simulated cardiac arrests. Team leaders are randomly designated. Designated teamleaders are instructed to lead their team from the position of the patient's head or remote from the patient.

DETAILED DESCRIPTION:
participants: physicians taking part in voluntary simulator-based workshops. Teams of 3-4 are formed. One teammember is randomly allocated as teamleader design: prospective, randomized, single-blind, cross-over intervention: teamleaders are randomized and instructed to lead their team from the conventional position at the patient's head or from a remote hands-off position data analysis: will be performed from videorecordings

ELIGIBILITY:
Inclusion Criteria:

* Physicians taking part in voluntary workshops

Exclusion Criteria:

* refusal to participate and/or being videorecorded

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Quantity of leadership | 5 minutes
  Number of leadership utterances made as defined by the adapted Leadership Behaviour Description Questionnaire

SECONDARY OUTCOMES:
Hands-on time | 5 minutes
  Hands-on time during the first 5 minutes of the cardiac arrest
Quality of leadership | 5 minutes
  Type of leadership utterances made as defined by the adapted Leadership Behaviour Description Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Marsch, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No
Secondary data can be changed Videorecordings of simulations are strictly confidential and cannot be shared